CLINICAL TRIAL: NCT02338401
Title: Effect of Fish Oil Supplementation on Resting Energy Expenditure, Skeletal Muscle Membrane Composition and Metabolism in Elderly Subjects.
Brief Title: Fish Oil Supplementation, Resting Energy Expenditure, Skeletal Muscle Membrane Composition and Metabolism in Elderly Subjects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Lawrence Spriet, Professor and Chair Human Health and Nutritional Sciences, University of Guelph
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: University of Guelph
Record Dates: First submitted 2015-01-10; First posted 2015-01-14 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Whole Body and Skeletal Muscle Energy Metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 Complete (Experimental): Oral ingestion of 3000 mg (5 capsules) of Omega-3 Complete (Jamieson Laboratories Ltd., Windsor, Ontario, Canada) per day for 12 weeks.
  Interventions: Dietary Supplement: Omega-3 Complete
- Placebo Pill (Placebo Comparator): Oral ingestion of 3 capsules of a placebo olive oil pill (Swanson Health Products, PO Box 2803 - Fargo, ND 58108 USA) per day for 12 weeks.
  Interventions: Dietary Supplement: Placebo Pill

INTERVENTIONS:
Dietary Supplement: Omega-3 Complete — Fish Oil Capsules
  Arms: Omega-3 Complete
Dietary Supplement: Placebo Pill — Olive Oil Capsules
  Arms: Placebo Pill

SUMMARY:
Resting metabolic rate (RMR) declines by 1-2% per decade after 20 years of age. This reduction is linked to a decrease in fat free mass (FFM) (10-20%) and the rate of energy expenditure of tissues (Manini 2010).

It has also been shown that as we age there is a:

* Concomitant reduction in basal fat and carbohydrate oxidation, most likely due to the decrease in RMR than to a change in respiratory exchange ratio (RER) (St-Onge and Gallagher 2010).
* A change towards a more saturated membrane of different tissues (Rabini et al 2002).

Incorporation of omega-3s, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), into cell membranes may alter energy metabolism by:

* Increasing the rate at which proteins operate (Hulbert 2007).
* Promoting the release of EPA and DHA into the cytosol which will act as ligands for peroxisome proliferator-activated receptors (PPARs) (Calder 2011). PPARs play an important role in energy homeostasis by regulating genes involved in lipid metabolism (Kota et al 2005).
* Augmenting protein synthesis through activation of the mTOR-p70s6k pathway (Di Girolamo et al 2014).

Supplementation with fish oil in older males and females:

* Increases whole muscle phospholipid profile of EPA and DHA (Smith et al 2011).
* Increases lean body mass (LBM), RMR, and fatty acid oxidation (Logan et al unpublished)
* Decreases carbohydrate oxidation (Logan et al unplubished). Skeletal muscle (SM) accounts for 20-30% of RMR (Zurlo et al 1990, Manini 2010), therefore it is tempting to speculate that these changes may occur by some of the mechanisms described earlier, with skeletal muscle being an important contributor.

To date there are no studies that have examined the effect of n-3 supplementation (3g/day)* on plasma membrane fatty acid composition, RMR and substrate oxidation, and the possible mechanisms behind it.

Therefore the purpose of this study is to determine whether in older adults (female and male), supplementation with n-3 alters:

1. RMR and fatty acid oxidation.
2. Membrane composition of whole muscle and sarcolemma.
3. Content of skeletal muscle membrane fatty acid transport proteins.
4. Dose response of NaKATPase and SERCA efficiency
5. Content of mitochondrial proteins
6. Expression and content of PPARs and proteins involved in translocation of FA transporters (AMPK, ERK1/2, CamKII).
7. Phosphorylation of AMPKα(THR172), ERK1/2(THR202 TYR204) and CaMKII(THR286).
8. Proteomic profile of skeletal muscle.
9. Body composition

ELIGIBILITY:
Inclusion Criteria:

* Between 60 and 75 years old
* Must currently practice a consistent diet and exercise regimen, and maintain this throughout the duration of the study

Exclusion Criteria:

* Have any medical condition (no evidence of significant cardiovascular disease or organ dysfunction, including hypertension, dyslipidemia, and diabetes mellitus), and hospitalization or surgeries
* Consume more than two meals of fish/wk and/or have taken an omega-3 supplement during the prior three months.
* Have a BMI > 30 kg/m2

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in skeletal muscle whole muscle membrane fatty acid composition from baseline | Baseline and 12 weeks
Change in skeletal muscle sodium pump (Na/K ATPase) activity (umol/mg protein/hour) | Baseline and 12 weeks
Change in skeletal muscle sarcoplasmic reticulum calcium (SERCA) ATPase activity (umol/mg protein/hour) | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change in whole body resting metabolic rate | Baseline, 6 and 12 weeks
Change in skeletal muscle membrane fatty acid transporter content | Baseline and 12 weeks
Change in skeletal muscle content of mitochondrial proteins | Baseline and 12 weeks
Change in skeletal muscle phosphorylation of AMPKα(THR172), ERK1/2(THR202 TYR204) and CaMKII(THR286) | Baseline and 12 weeks
Change in skeletal muscle PPARs content | Baseline and 12 weeks
Change in body composition | Baseline, 6 and 12 weeks

OTHER OUTCOMES:
Change in Whole Body Resting Fat Oxidation From Baseline | Baseline, 6 and 12 weeks
Change in Whole Body Resting Carbohydrate Oxidation From Baseline | Baseline, 6 and 12 weeks
Change in Fasted Blood Triglyceride Concentration From Baseline | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph, Guelph, Ontario, Canada